CLINICAL TRIAL: NCT06436703
Title: A STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF MODIFIED RNA VACCINES AGAINST INFLUENZA IN HEALTHY ADULTS
Brief Title: A Study About Modified RNA Vaccines Against Influenza in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C4781013; NCT06436703 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-05-24; First posted 2024-05-31 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study will be an observer-blinded and Sponsor-unblinded study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (19):
- SSA: Influenza ModRNA Vaccine 2A (Experimental): - Single Dose on Day 1
  Interventions: Biological: Influenza ModRNA Vaccine
- SSA: Influenza ModRNA Vaccine 3A (Experimental): - Single Dose on Day 1
  Interventions: Biological: Influenza ModRNA Vaccine
- SSA: Influenza ModRNA Vaccine 4A (Experimental): - Single Dose on Day 1
  Interventions: Biological: Influenza ModRNA Vaccine
- SSA: Influenza ModRNA Vaccine 5A (Experimental): - Single dose on Day 1
  Interventions: Biological: Influenza ModRNA Vaccine
- SSA: QIV1 (Active Comparator): - Single dose on Day 1
  Interventions: Biological: Quadrivalent Influenza Vaccine (QIV)
- SSB: Influenza ModRNA Vaccine 3B (Experimental): - Single Dose on Day 1
  Interventions: Biological: Influenza ModRNA Vaccine
- SSB: Influenza ModRNA Vaccine 4B (Experimental): - Single Dose on Day 1
  Interventions: Biological: Influenza ModRNA Vaccine
- SSB: Influenza ModRNA Vaccine 5B (Experimental): - Single dose on Day 1
  Interventions: Biological: Influenza ModRNA Vaccine
- SSB: QIV2 (Active Comparator): - Single Dose on Day 1
  Interventions: Biological: Quadrivalent Influenza Vaccine (QIV)
- SSB: QIV3 (Active Comparator): - Single Dose on Day 1
  Interventions: Biological: Quadrivalent Influenza Vaccine (QIV)
- SSC: Influenza ModRNA Vaccine 3C (Experimental): - Single Dose on Day 1
  Interventions: Biological: Influenza ModRNA Vaccine
- SSC: Influenza ModRNA Vaccine 4C (Experimental): - Single Dose on Day 1
  Interventions: Biological: Influenza ModRNA Vaccine
- SSC: Influenza ModRNA Vaccine 5C (Experimental): - Single Dose on Day 1
  Interventions: Biological: Influenza ModRNA Vaccine
- SSC: Influenza ModRNA Vaccine 6C (Experimental): - Single Dose on Day 1
  Interventions: Biological: Influenza ModRNA Vaccine
- SSC: Influenza ModRNA Vaccine 7C (Experimental): - Single Dose on Day 1
  Interventions: Biological: Influenza ModRNA Vaccine
- SSC: Influenza ModRNA Vaccine 8C (Experimental): - Single Dose on Day 1
  Interventions: Biological: Influenza ModRNA Vaccine
- SSC: Influenza ModRNA Vaccine 9C (Experimental): - Single dose on Day 1
  Interventions: Biological: Influenza ModRNA Vaccine
- SSC: QIV2 (Active Comparator): - Single Dose on Day 1
  Interventions: Biological: Quadrivalent Influenza Vaccine (QIV)
- SSC: QIV3 (Active Comparator): - Single Dose on Day 1
  Interventions: Biological: Quadrivalent Influenza Vaccine (QIV)

INTERVENTIONS:
Biological: Influenza ModRNA Vaccine — Intramuscular injection
  Arms: SSA: Influenza ModRNA Vaccine 2A; SSA: Influenza ModRNA Vaccine 3A; SSA: Influenza ModRNA Vaccine 4A; SSA: Influenza ModRNA Vaccine 5A; SSB: Influenza ModRNA Vaccine 3B; SSB: Influenza ModRNA Vaccine 4B; SSB: Influenza ModRNA Vaccine 5B; SSC: Influenza ModRNA Vaccine 3C; SSC: Influenza ModRNA Vaccine 4C; SSC: Influenza ModRNA Vaccine 5C; SSC: Influenza ModRNA Vaccine 6C; SSC: Influenza ModRNA Vaccine 7C; SSC: Influenza ModRNA Vaccine 8C; SSC: Influenza ModRNA Vaccine 9C
Biological: Quadrivalent Influenza Vaccine (QIV) — Intramuscular injection
  Arms: SSA: QIV1; SSB: QIV2; SSB: QIV3; SSC: QIV2; SSC: QIV3

SUMMARY:
The purpose of this study is to learn if modified RNA (modRNA) vaccines for the prevention of influenza are:

* safe; and
* how these vaccines produce an immune response in generally healthy adults. Immune response is the way the body protects itself against things it sees as harmful or foreign.

RNA (also called ribonucleic acid) is one of two types of nucleic acid made by cells. RNA contains information that has been copied from DNA (the other type of nucleic acid). Cells make several different forms of RNA, and each form has a specific job in the cell. Many forms of RNA have functions related to making proteins. RNA is also the genetic material of some viruses instead of DNA. RNA can be made in the laboratory and used in research studies. Also called ribonucleic acid.

Influenza is term used for flu illness. It is an infection caused by a virus that affects your mouth, nose, and throat.

The study is seeking for participants who:

* are at least 18 years of age
* have not received an influenza vaccine within the last 6 months
* are generally healthy

This study will be divided into three sub-studies: Substudy A (SSA), Substudy B (SSB), and Substudy C (SSC).

All participants, regardless of sub-study, will receive 1 dose of either of the following vaccines as an injection into their arm:

* 1 of the modRNA influenza vaccines that is being studied; or
* an approved influenza vaccine approved for use in their respective age group.

Participants will be involved in this study for about 6 months. During this time, participants will have at least 3 clinic visits.

ELIGIBILITY:
Key Inclusion Criteria

Applies to all 3 substudies:

* participants ≥18 years of age.
* generally healthy participants.

Substudy C ONLY:

- receipt of licensed influenza vaccination for the 2023-2024 flu season at least 6 months ago.

Key Exclusion Criteria

All 3 substudies:

* diagnosis of influenza (by clinical testing) in the last 6 months.
* immunocompromised individuals with known or suspected immunodeficiency
* receipt of any investigational or licensed influenza vaccines within 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1202 (Actual)
Dates: Start 2024-05-23 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
SSA - Percentage of Participants Reporting Local Reactions After Vaccination | From Day 1 Through at least Day 7 After Vaccination
  Pain at the injection site, redness, and swelling.
SSA - Percentage of Participants Reporting Systemic Events After Vaccination | From Day 1 Through at least Day 7 After Vaccination
  Fever, fatigue, headache, chills, vomiting, diarrhea, new or worsened muscle pain, and new or worsened joint pain.
SSA - Percentage of Participants Reporting Adverse Events After Vaccination | From Day 1 Through 4 Weeks After Vaccination
  As elicited by investigational site staff
SSA - Percentage of Participants Reporting Serious Adverse Events (SAE) | From Day 1 Through 6 Months After Vaccination
  As elicited by investigational site staff
SSA - Percentage of Participants Reporting Newly Diagnosed Chronic Medical Conditions (NDCMCs) | From Day 1 Through 6 Months After Vaccination
  As elicited by investigational site staff
SSA - Percentage of Participants Reporting Medically Attended AEs (MAEs) | From Day 1 Through 6 Months After Vaccination
  As elicited by investigational site staff
SSB - Percentage of Participants Reporting Local Reactions After Vaccination | From Day 1 Through at least Day 7 After Vaccination
  Pain at injection site, redness, and swelling.
SSB - Percentage of Participants Reporting Systemic Events After Vaccination | From Day 1 Through at least Day 7 After Vaccination
  Fever, fatigue, headache, chills, vomiting, diarrhea, new or worsened muscle pain, and new or worsened joint pain.
SSB - Percentage of Participants Reporting Adverse Events After Vaccination | From Day 1 Through 4 Weeks After Vaccination
  As elicited by investigational site staff
SSB - Percentage of Participants Reporting Serious Adverse Events (SAE) | From Day 1 Through 6 Months After Vaccination
  As elicited by investigational site staff
SSB - Percentage of Participants Reporting Newly Diagnosed Chronic Medical Conditions (NDCMCs) | From Day 1 Through 6 Months After Vaccination
  As elicited by investigational site staff
SSB - Percentage of Participants Reporting Medically Attended AEs (MAEs) | From Day 1 Through 6 Months After Vaccination
  As elicited by investigational site staff
SSC - Percentage of Participants Reporting Local Reactions After Vaccination | From Day 1 Through at least Day 7 After Vaccination
  Pain at the injection site, redness, and swelling.
SSC - Percentage of Participants Reporting Systemic Events After Vaccination | From Day 1 Through at least Day 7 After Vaccination
  Fever, fatigue, headache, chills, vomiting, diarrhea, new or worsened muscle pain, and new or worsened joint pain.
SSC - Percentage of Participants Reporting Adverse Events After Vaccination | From Day 1 Through 4 Weeks After Vaccination
  As elicited by investigational site staff
SSC - Percentage of Participants Reporting Serious Adverse Events (SAE) | From Day 1 Through 6 Months After Vaccination
  As elicited by investigational site staff
SSC - Percentage of Participants Reporting Newly Diagnosed Chronic Medical Conditions (NDCMCs) | From Day 1 Through 6 Months After Vaccination
  As elicited by investigational site staff
SSC - Percentage of Participants Reporting Medically Attended AEs (MAEs) | From Day 1 Through 6 Months After Vaccination
  As elicited by investigational site staff

SECONDARY OUTCOMES:
SSA - HAI Geometric Mean Titers (GMTs) for each strain | 4 Weeks After Vaccination
  As measured at the central laboratory
SSA - HAI geometric mean fold rise (GMFR) for each strain | 4 Weeks After Vaccination
  As measured at the central laboratory
SSA - The proportion of participants achieving HAI seroconversion for each strain | 4 Weeks After Vaccination
  As measured at the central laboratory
SSA - The proportion of participants with HAI titers ≥1:40 for each strain | Baseline and 4 Weeks After Vaccination
  As measured at the central laboratory
SSB - HAI geometric mean titers (GMTs) for each strain | 4 Weeks After Vaccination
  As measured at the central laboratory
SSB - HAI geometric mean fold rise (GMFR) for each strain | 4 Weeks After Vaccination
  As measured at the central laboratory
SSB - The proportion of participants achieving HAI seroconversion for each strain | 4 Weeks After Vaccination
  As measured at the central laboratory
SSB - The proportion of participants with HAI titers ≥1:40 for each strain | Baseline and 4 Weeks After Vaccination
  As measured at the central laboratory

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (32):
- United States (32):
  - Alliance for Multispecialty Research, LLC, Mobile, Alabama
  - Headlands Research - Scottsdale, Scottsdale, Arizona
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Orange County Research Center, Lake Forest, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Clinical Research Consulting, Milford, Connecticut
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - Research Centers of America ( Hollywood ), Hollywood, Florida
  - Research Centers of America, Hollywood, Florida
  - Palm Springs Community Health Center, Miami Lakes, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Headlands Research Orlando, Orlando, Florida
  - Qps-Mra, Llc, South Miami, Florida
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Alliance for Multispecialty Research, LLC, New Orleans, Louisiana
  - Prism Research LLC dba Nucleus Network, Saint Paul, Minnesota
  - Clinical Research Professionals, Chesterfield, Missouri
  - Alliance for Multispecialty Research, LLC, Kansas City, Missouri
  - Rochester Clinical Research, LLC, Rochester, New York
  - Duke Vaccine and Trials Unit, Durham, North Carolina
  - M3 Wake Research, Inc., Raleigh, North Carolina
  - DM Clinical Research - Philadelphia, Philadelphia, Pennsylvania
  - Headlands Horizons LLC, Brownsville, Texas
  - SMS Clinical Research, Mesquite, Texas
  - Clinical Trials of Texas, LLC dba Flourish Research, San Antonio, Texas
  - Clinical Trials of Texas, LLC, San Antonio, Texas
  - Dynamed Clinical Research, LP d/b/a DM Clinical Research, Tomball, Texas
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Alliance for Multispecialty Research, LLC, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4781013